CLINICAL TRIAL: NCT01485263
Title: Analysis of Visual-Motor Task Electrophysiological Activity During Deep Brain Stimulation for Treatment-Resistant Movement Disorders
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: George Washington University (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110157; 11-N-0157
Record Dates: First submitted 2011-12-02; First posted 2011-12-05 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07-06

CONDITIONS: Obsessive-Complusive Disorder
Keywords: Deep Brain Stimulation; OCD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Objective

The objective of this pilot study is to characterize the abnormal neuronal firing patterns of basal ganglia neurons and those in the premotor cortex in patients with treatment-resistant movement disorders undergoing deep brain stimulation (DBS) surgery.

Study population

Fifteen adult patients with treatment-resistant movement disorders who are undergoing deep brain stimulation surgery at Suburban Hospital, Bethesda, Maryland, will be studied.

Design

This is a physiology study of treatment-resistant movement disorder patients who have been scheduled for implantation of a deep brain stimulation device into the Nucleus accumbens. Prior to surgery, patients will learn a rewarded visual-motor task and undergo magnetoencephalography. The task will be repeated during DBS surgery, with collection of information on electrical activity including single neuronal unit and local field potentials. The task and MEG will be repeated 3-4 months after surgery. The collected data will be analyzed for coherence patterns during rest and rewarded movements.

Outcome measures

We plan to characterize and quantify the oscillatory activity present in motor circuits of treatment-resistant movement disorder patients during rewarded visually guided movements. We hypothesize that during visually guided movements, neuronal coherence will be significantly increased relative to resting periods. Thus, by better understanding the alteration in oscillatory patterns in these patients, we hope to develop better DBS stimulation paradigms in order to better treat this disease in the future.

DETAILED DESCRIPTION:
Objective:

The objective of this pilot study is to characterize the abnormal neuronal firing patterns of basal ganglia and thalamic neurons and those in the premotor cortex in patients with treatment-resistant movement disorders undergoing deep brain stimulation (DBS) surgery. Neuronal activity will be studied in a decision-making task guided by reward. Secondary objectives will involve study of how activity in the brain is modulated in such a task and how DBS can influence the cerebral activity related to decision-making.

Study population:

Fifteen adult patients with treatment-resistant movement disorders (Essential tremor or Parkinson s disease) who are undergoing deep brain stimulation surgery at Suburban Hospital, Bethesda, Maryland, will be studied.

Design:

This is a physiology study of medically refractory patients who have been scheduled for implantation of a deep brain stimulation device into basal ganglia or thalamic structures. Prior to surgery, patients will learn a rewarded visual-motor task and undergo magnetoencephalography (MEG). The task will be repeated during DBS surgery, with collection of information on electrical activity including single neuronal unit and local field potentials. The task and MEG will be repeated 3 and 6 months after surgery.

Outcome measures:

The collected data will be analyzed for coherence patterns during rest and rewarded movements. We plan to characterize and quantify the oscillatory activity present in motor circuits of patients during rewarded visually guided movements. We hypothesize that during visually guided movements, neuronal coherence will be significantly increased relative to resting periods. Activity during surgery will be compared with MEG recordings in the same task both before and after surgery. By understanding the alteration in oscillatory patterns in these patients, we hope to improve DBS stimulation paradigms in order to optimize treatment protocols.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult patients (over 18 years of age) with severe treatment-resistant ET or PD who are scheduled for deep brain stimulation surgery at Suburban Hospital

Able to provide Informed Consent

EXCLUSION CRITERIA:

Subjects who are not willing or able to safely tolerate the study procedures

Subjects who have untreated depression or psychiatric disorder

Subjects who use illicit substances

Subjects who are pregnant

Subjects who are claustrophobic

Subjects who have metallic dental fillings.

Subjects who have any of the following: cardiac pacemaker; implanted cardiac defibrillator; aneurysm clip; neuro or bone stimulator; insulin or infusion pump; implanted drug infusion device; cochlear, otologic, or ear implant; prostate radiation seeds; IUD (intrauterine device); transdermal medication patch (Nitro); any type of prosthesis (eye, penile); heart valve prosthesis; shunt (spinal/intraventricular); wire sutures or surgical staples; bone/joint pin, screw, nail, plate; body tattoos or makeup (eyeliner/lip); body piercing(s) (non-removable); breast tissue expander; any metallic implants or objects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05-26; Study Completion 2017-07-06

PRIMARY OUTCOMES:
The primary objective of this trial is to evaluate and quantify neuronal coherence in basal ganglia structures at rest and during rewarded movement.

SECONDARY OUTCOMES:
The latency and amplitude of evoked activity related to decision-making processing. We will also measure the reaction times and the number of errors.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)

REFERENCES:
- [Background] Alexander GE, DeLong MR, Strick PL. Parallel organization of functionally segregated circuits linking basal ganglia and cortex. Annu Rev Neurosci. 1986;9:357-81. doi: 10.1146/annurev.ne.09.030186.002041. No abstract available. PMID 3085570
- [Background] Alexander GE, Crutcher MD. Functional architecture of basal ganglia circuits: neural substrates of parallel processing. Trends Neurosci. 1990 Jul;13(7):266-71. doi: 10.1016/0166-2236(90)90107-l. PMID 1695401
- [Background] Alexander GE, Crutcher MD. Preparation for movement: neural representations of intended direction in three motor areas of the monkey. J Neurophysiol. 1990 Jul;64(1):133-50. doi: 10.1152/jn.1990.64.1.133. PMID 2388061